CLINICAL TRIAL: NCT02327091
Title: Phase 3 Study of Vitamin D Analog (Alfacalcidol) on Muscle Strength in Elderly Indonesian Women Who Have Low Handgrip Strength
Brief Title: The Effect of Alfacalcidol on Muscle Strength in Elderly Indonesian Women : A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Anugrahini, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 269/PT02.FK
Record Dates: First submitted 2013-01-28; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Muscle Weakness
Keywords: Alfacalcidol; Falls; Handgrip; Muscle strength; Sarcopenia
MeSH Terms: conditions — Muscle Weakness; Sarcopenia | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- white rice flour capsule (Placebo Comparator): One group of 47 subjects received alfacalcidol 0.5 mcg/day and the other group received placebo for 12 weeks
- alfacalcidol (Active Comparator): One group of 47 subjects received alfacalcidol 0.5 mcg/day and the other group received placebo
  Interventions: Drug: alfacalcidol

INTERVENTIONS:
Drug: alfacalcidol — One group of 47 subjects received alfacalcidol 0.5 mcg/day and the other group received placebo
  Other Names: BoneOne, C27H4402
  Arms: alfacalcidol

SUMMARY:
The age-related increase in falls is strongly associated with a decline in muscle strength by the mechanism of sarcopenia. There has been great interest in developing approaches to counteract the effects of sarcopenia, and thereby reduce the age-related decline in muscle mass with vitamin D that have muscular effect. However, a limited number of studies demonstrate a vitamin D analog (alfacalcidol) increase in lower body muscle strength in adults with vitamin D deficiency. A double-blinded randomized controlled trial was conducted in order to determine the effect of alfacalcidol on the upper-body muscle strength in Indonesian elderly women in age group of 60 or more who had low handgrip strength.

DETAILED DESCRIPTION:
A total 122 elderly women were enrolled to this study. It was determined subjects with handgrip strength less than 22 kg and measured using handheld dynamometer. There were 95 subjects fulfilled the eligible criteria. These subjects were randomized into two groups, one group of 47 subjects received alfacalcidol 0.5 mcg/day and the other group received placebo. Each subject was given calcium 500 mg/day. After 12 weeks of intervention, 88 subjects had the second muscle strength measurement (7 dropped out).

ELIGIBILITY:
Inclusion Criteria:

* Elderly women in age group of 60 or more
* Subjects with handgrip strength less than or equal to 22 kg

Exclusion Criteria:

* Hypercalcemia (serum calcium > 10.5 mg / dL)
* Can not understand instructions well (MMSE scale < 16)
* Depression (Geriatric Depression Scale> 10)
* Fracture, deformity, and pain with a visual analog scale (VAS) ≥ 4 on fingers and joints of the upper limb when the examination will be conducted
* Heart failure fc. III-IV or uncontrolled according to the New York Heart Association (NYHA)
* Neurological conditions (epilepsy, acute stroke, Parkinson's)
* Malignant hypertension (systolic blood pressure ≥ 200 mmHg and or diastolic blood pressure ≥ 120 mmHg)
* Blood malignancies and solid tumors
* Decreased function of the liver (cirrhosis, ALT increase above 2 times the upper normal limit )
* Refusing to follow the research / not willing controls

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement of muscle strength in the group that received alfacalcidol compared to placebo | 12 weeks
  After 12 weeks of intervention, 88 subjects had the second muscle strength measurement

CONTACTS AND LOCATIONS:
Overall Officials: Iin Anugrahini, Principal Investigator — Internal of Medicine, University of Indonesia
Locations (1):
- Division of Geriatrics, Department of Internal Medicine, University of Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia